CLINICAL TRIAL: NCT03371563
Title: Clinical Course, Serologic Response and Long-term Outcome in Elderly Patients With Early Lyme Borreliosis
Brief Title: Erythema Migrans in Elderly
Status: Completed | Type: Observational
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Daša Stupica, MD, PhD, University Medical Centre Ljubljana
Other Study IDs: EM-elderly
Record Dates: First submitted 2017-12-08; First posted 2017-12-13 (Actual); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Lyme Disease; Erythema Migrans; Elderly Infection
MeSH Terms: conditions — Lyme Disease; Glossitis, Benign Migratory | interventions — Anti-Bacterial Agents

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- elderly patients
  Interventions: Drug: Antibiotics
- middle-aged patients
  Interventions: Drug: Antibiotics
- controls
  Interventions: Other: no intervention
- young patients
  Interventions: Drug: Antibiotics

INTERVENTIONS:
Drug: Antibiotics — Patients were treated with antibiotics for Lyme disease.
  Groups: elderly patients; middle-aged patients; young patients
Other: no intervention — controls were not given antibiotics
  Groups: controls

SUMMARY:
The investigators will focus on elderly patients with early Lyme borreliosis with the aim of assessing clinical course, serological response and treatment outcome of the disease as compared to younger adults. Furthermore, the investigators will compare the prevalence of nonspecific symptoms among patients and among age-matched controls without a history of Lyme borreliosis.

ELIGIBILITY:
Inclusion Criteria:

* erythema migrans

Exclusion Criteria:

* pregnancy or lactation
* immunocompromised
* taking antibiotic with antiborrelial activity within 10 days
* received <10 days of antibiotic therapy for erythema migrans
* had an intercurrent episode of Lyme borreliosis during follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: young (18-44 years), middle-aged (45-64 years) and elderly 65 or more years) patients with erythema migrans
Sampling Method: Non-Probability Sample
Enrollment: 1220 (Actual)
Dates: Start 2006-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Occurrence of objective clinical manifestations of Lyme borreliosis and post-Lyme symptoms at 14 days postenrollment in patients treated for erythema migrans | Study point: at 14 days post-enrollment.
  At follow-up at 14 days patients were examined physically and were asked an open question about health-related symptoms. Symptoms that had newly develop or worsened since the onset of the multiple erythema migrans and which will had no other known medical explanation were regarded as post-Lyme symptoms.
  Complete response to treatment will be defined as a return to pre-Lyme health status. Partial response will be defined as the presence of post-Lyme symptoms, while occurrence of new objective signs of Lyme borreliosis was interpreted as failure.
Occurrence of objective clinical manifestations of Lyme borreliosis and post-Lyme symptoms at 2 months postenrollment in patients treated for erythema migrans with doxycycline for 7 or 14 days | Study point: at 2 months post-enrollment.
  At follow-up at 2 months patients were examined physically and were asked an open question about health-related symptoms. Symptoms that hed newly develop or worsened since the onset of the erythema migrans and which will had no other known medical explanation were regarded as post-Lyme symptoms.
  Complete response to treatment was defined as a return to pre-Lyme health status. Partial response will be defined as the presence of post-Lyme symptoms, while occurrence of new objective signs of Lyme borreliosis, and/ or persistence of borreliae as detected by culture of skin re-biopsy sample, and/or persistence of erythema migrans at more than 2 months post-treatment was be interpreted as failure.
Occurrence of objective clinical manifestations of Lyme borreliosis and post-Lyme symptoms at 6 months postenrollment in patients treated for erythema migrans | Study point: at 6 months post-enrollment.
  At follow-up at 6 months patients were examined physically and were asked an open question about health-related symptoms. Symptoms that had newly develop or worsened since the onset of the erythema migrans and which had no other known medical explanation were regarded as post-Lyme symptoms. Complete response to treatment was defined as a return to pre-Lyme health status. Partial response was defined as the presence of post-Lyme symptoms, while occurrence of new objective signs of Lyme borreliosis, and/ or persistence of borreliae as detected by culture of skin re-biopsy sample, and/or persistence of erythema migrans at more than 2 months post-treatment was interpreted as failure.
Occurrence of objective clinical manifestations of Lyme borreliosis and post-Lyme symptoms at 12 months postenrollment in patients treated for erythema migrans | Study point: at 12 months post-enrollment.
  At 12 months patients were examined physically and were asked an open question about health-related symptoms.
  Symptoms that had develop or worsened since the onset of the erythema migrans and which had no other known medical explanation were regarded as post-Lyme symptoms. Complete response to treatment was defined as a return to pre-Lyme health status. Partial response was defined as the presence of post-Lyme symptoms, while occurrence of new objective signs of Lyme borreliosis, and/ or persistence of borreliae as detected by culture of skin re-biopsy sample, and/or persistence of erythema migrans at more than 2 months post-treatment was interpreted as failure.

SECONDARY OUTCOMES:
Change in occurrence of nonspecific symptoms from baseline to 6 months and to 12 months post-enrollment in patients with erythema migrans and control subjects | Study points will be: at enrollment, at 6, and at 12 months post-enrollment
  Patients completed a written questionnaire asking whether they had had any of 8 nonspecific symptoms (fatigue, arthralgias, headache, myalgias, paresthesias, memory difficulties, concentration difficulties, irritability) within the preceding week. Control subjects completed the same 8-symptom questionnaire as the patients within 14 days of the examination date of the corresponding patient at enrollment, and again at 6 and 12 months. Patients and controls graded the severity of each individual symptom on a 10-cm visual analogue scale (10 = most severe).

IPD SHARING:
Plan to Share IPD: Undecided